CLINICAL TRIAL: NCT07128420
Title: Microneedle Treatment of Chronic Phase Peyronie's Disease: A Pilot Clinical Trial
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Luke Witherspoon, Urologist, Ottawa Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20250265-01H
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Peyronie's Disease
Keywords: Peyronie's disease; Microneedle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Microneedle application to Peyronie's plaque tissue (Experimental)
  Interventions: Device: Application of 3 sessions of microneedle therapy

INTERVENTIONS:
Device: Application of 3 sessions of microneedle therapy — Enrolled study participants will receive 3-4 treatments of microneedling to the affected area.
  Study participants will microneedling (Fusion Tip Potenza Fractional Radiofrequency Microneedle Electrosurgical Unit, Jeisys Medical Inc, Seoul, KR) at a depth of 2.0 to 2.75mm.

SUMMARY:
Peyronie's Disease (PD) is a disorder of the penis where scar tissue (composed of excessive and disorganized collagen) known as a "plaque," forms along the shaft of the penis. This plaque can lead to permanent penile deformity (curvature, narrowing, indentation, hinging), loss of penile length, erectile dysfunction, and pain during intercourse. Research has shown PD to negatively impact the quality of life and cause significant psychosocial distress for many men.

This study proposes the use of microneedle treatment of chronic phase PD. Microneedling is a minimally invasive technique that creates tiny injuries in scarred tissues, which encourages a controlled healing process.

This will be a pilot clinical trial evaluating the safety and feasibility of using microneedling treatment in the management of chronic phase PD. Enrolled study participants will undergo an initial clinical assessment of their PD which involves penile measurements at flaccid and erect states, a curvature assessment with duplex ultrasound, and will be asked to complete the International Index of Erectile Function Questionnaire (IIEF-5), and Peyronie's Disease Questionnaire (PDQ). They will then undergo 3-4 treatment sessions at 6-8 week intervals. This will then be followed by a short and long-term follow-up at 24 and 52-54 weeks, respectively.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy males aged 18 or older in a stable relationship with a female partner/spouse (for at least 3 months and willing to have vaginal intercourse with their female partner/spouse).Non heterosexual men are also included; however they need not fill out the PDQ questionnaire as it pertains to those having intercourse with females.

  2. Diagnosis of PD for at least 12 months with evidence of stable disease as determined by the investigator (i.e. no change in penile curve for at least 6 months and absence of pain).

  3. Penile curvature of 30º-90º in the dorsal, lateral, or dorsal/lateral plane (must be possible to delineate the single plane of maximal curvature for evaluation)

  4. Signed informed IRB-approved consent agreement; signed authorization form to allow disclosure of protected information.

  5. Ability to read, complete, and understand the various rating instruments in English.

Exclusion Criteria:

* 1. Penile curvature of <30º or >90º

  2. Any conditions affecting the penis such as a chordee in the presence or absence of hypospadias; thrombosis of the dorsal penile artery; infiltration by a benign or malignant mass or an infectious agent; ventral curvature from any cause; presence of an active sexually transmitted disease.

  3. Failure to achieve a sufficient 8/10 erection (after prostaglandin E or Trimix administration), in the opinion of the investigator, to accurately measure the penile deformity.

  4. Calcified plaque as evident by appropriate radiographic evaluation, i.e., penile ultrasound that would prevent treatment with microneedling.

  5. Isolated hourglass deformity of the penis without curvature

  6. Treatment or plans to undergo treatment for PD, including but not limited to any previous surgery, oral/topical agents within 3 months, intralesional medical therapies within 3 months, extracorporeal shock wave therapy within 6 months, or use of mechanical devices within 2 weeks before the start of the study

  7. Use of or plans to use a mechanical device to induce a passive erection within 2 weeks before the start of study.

  8. Erectile Dysfunction that was unresponsive to PDE5 inhibitors

  9. Received an investigation drug or treatment within 30 days before start of the study.

  10. At any time, received collagenase clostridium histolyticum (CCH) for the treatment of PD.

  11. Currently on anti-coagulation medications.

  12. History of HSV

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Safety | 52 weeks
  Given that this is a pilot study, safety is a critical outcome alongside feasibility and efficacy. Adverse events (AEs) and serious adverse events (SAEs) related to microneedling will be collected, documented, and analyzed to evaluate the safety profile of the intervention. AEs will be assessed at every treatment and follow-up visit through direct questioning, physical examinations, and spontaneous participant reports. Investigators will use a standardized adverse event log to capture the nature, severity, duration, frequency, and outcome of all events.
  The incidence of AEs and SAEs will be summarized descriptively using counts and percentages. Events will be categorized by severity (mild, moderate, severe), expectedness (anticipated vs. unanticipated), and relationship to the intervention (definitely, probably, possibly, unlikely, unrelated).

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided